CLINICAL TRIAL: NCT03400852
Title: A Multicenter, Randomized, Parallel Group, Double Blind, Multiple Dose, Placebo Controlled Study to Assess the Efficacy and Safety of MNK-1411 in Male Participants 4 to 8 Years of Age With Duchenne Muscular Dystrophy
Brief Title: A Study to Assess the Efficacy and Safety of MNK-1411 in Duchenne Muscular Dystrophy
Acronym: BRAVE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Mallinckrodt ARD LLC (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNK14112096; 2017-004139-35 (EudraCT Number)
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Muscular Dystrophy; DMD; Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies | interventions — Cosyntropin

STUDY DESIGN:
Intervention Model Description: In the double-blind period, participants are randomized to receive study drug or placebo. It is followed by an open label period wherein all participants receive study drug.
Who Masked: Participant, Investigator
Masking Description: Double blind (Investigator/Participant) The Care Provider and Outcomes Assessor were also blinded, but it is a double-blind trial, followed by an open-label period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Period 1: MNK-1411 (Experimental): Participants receive MNK-1411 at a dosing volume appropriate to body weight during Period 1
  Interventions: Drug: MNK-1411
- Period 1: Placebo (Experimental): Participants receive placebo at a volume appropriate to body weight during Period 1
  Interventions: Other: Placebo
- Period 2: MNK-1411 (Experimental): All participants receive MNK-1411 at a dosing volume appropriate to body weight during Period 2
  Interventions: Drug: MNK-1411

INTERVENTIONS:
Drug: MNK-1411 — MNK-1411 (1 mg/mL suspension) for subcutaneous injection
  Other Names: Cosyntropin acetate; Tetracosactide Hexaacetate
  Arms: Period 1: MNK-1411; Period 2: MNK-1411
Other: Placebo — Placebo suspension for subcutaneous injection
  Other Names: Matching Placebo
  Arms: Period 1: Placebo

SUMMARY:
This is a multicenter, double blind, placebo controlled, multiple dose study to examine the safety and efficacy of MNK-1411 in male subjects 4 to 8 years of age (inclusive) with Duchenne Muscular Dystrophy (DMD).

DETAILED DESCRIPTION:
The main purpose of this study is to determine the effect of MNK-1411 on motor function in participants with Duchenne Muscular Dystrophy (DMD). Information is collected only from caretakers who are fluent in English, using the Pediatric Outcomes Data Collection Instrument (PODCI).

The PODCI is a validated 86-question instrument completed by the parent or legal guardian of children 2 to 10 years of age to assess a variety of health outcome measures (Uzark et al, 2012). This study will only collect information for the PODCI domains of sports and physical functioning and transfer/basic mobility.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a documented diagnosis of Duchenne Muscular Dystrophy (DMD) confirmed by complete dystrophin deficiency (by immunofluorescence and/or immunoblot), or identifiable mutation in the DMD gene where reading frame can be predicated as "out of frame," or complete dystrophin gene sequencing consistent with DMD; AND in the opinion of the Investigator, a typical clinical profile consistent with DMD.
2. Participants taking approved treatments for DMD (by a Health Authority) that target dystrophin gene mutations (e.g., eteplirsen or ataluren) may be enrolled in the study if they have been on a stable dose for 30 days prior to the first dose of study drug, and plan to remain on that dose throughout the study.

Exclusion Criteria:

1. Participant has had previous systemic treatment with corticosteroids within 2 months prior to the Screening Visit. Exception: In subjects who were down-titrated to a physiological dose of corticosteroids (ie, 3mg/m2 of prednisone or deflazacort) a maximum of 1 month of no greater than a physiological dose followed by 1 month completely off corticosteroids prior to the Screening Visit will be acceptable for study entry. Transient previous use of corticosteroids will be evaluated on a case-by-case basis by the sponsor or designee. The use of topical or intra-articular corticosteroids is permitted during the study
2. Participant is unable to complete the 10 meter Walk/Run test at the Screening and/or Baseline Visit.
3. Participant has Type 1 or Type 2 diabetes mellitus.
4. Participant has a history of chronic active hepatitis including acute or chronic hepatitis B, or acute or chronic hepatitis C.
5. Participant has a history of tuberculosis (TB) infection, any signs/symptoms of TB, or any close contact with an individual with an active TB infection.
6. Participant has known immune compromised status (not related to disease/condition under study), including but not limited to, individuals who have undergone organ transplantation or who are known to be positive for the human immunodeficiency virus.

Ages: 4 Years to 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Lead, Study Director — Mallinckrodt
Locations (16):
- United States (5):
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Monroe Carell Jr Childrens Hospital at Vanderbilt, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - UT Health Science Center, San Antonio, San Antonio, Texas
- University Multiprofile Hospital for Active Treatment Aleksandrovska EAD, Sofia, Bulgaria
- Edith Wolfson Medical Center, Holon, Israel
- Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy, Italy
- Mexico (3):
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Neurociencias Estudios Clinicos S.C., Culiacán, Sinaloa
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
- Clinic of Neurology and Psychiatry for Children and Youth, Belgrade, Serbia
- Spain (3):
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Sant Joan de Deu - PIN, Esplugues de Llobregat
  - Hospital Universitari i Politecnic La Fe Valencia, Valencia
- Mersin Universitesi Tip Fakultesi Hastanesi, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Discussion of statistical endpoints and analysis are included in manuscripts. Summary aggregate (basic) results (including adverse events information) and the study protocol are made available on clinicaltrials.gov (NCT03400852) when required by regulation. Individual de-identified patient data will not be disclosed. Requests for additional information should be directed to the company at medinfo@mnk.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four participants with Duchenne Muscular Dystrophy (DMD) who chose to discontinue the double-blind period prior to Week 24 entered the open label extension (OLE, Period 2). Participants who did not enter OLE Period were followed up to Week 28.
Pre-assignment Details: After screening, 44 participants from 8 countries were enrolled into Period 1
Period: Blinded Treatment Period
Arm/Group | Period 1: MNK-1411 | Period 1: Placebo | Period 2: MNK-1411
Started (Period 2 arm not included in Period 1) | 29 | 15 | 0
Completed | 20 | 9 | 0
Not Completed | 9 | 6 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Study terminated by sponsor | 8 | 4 | 0
Period: Open Label Period
Arm/Group | Period 1: MNK-1411 | Period 1: Placebo | Period 2: MNK-1411
Started (Period 1 arms not included in Period 2) | 0 | 0 | 24
Completed | 0 | 0 | 2
Not Completed | 0 | 0 | 22
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Study terminated by sponsor | 0 | 0 | 21

BASELINE CHARACTERISTICS:
Population: All participants enrolled into the study.
Groups:
- Period 1: MNK-1411: All participants who received any dose of MNK-1411 in Period 1
- Period 1: Placebo: All patients who received placebo in Period 1
- Total: Total of all reporting groups
Arm/Group | Period 1: MNK-1411 | Period 1: Placebo | Total
Number analyzed (Participants) | 29 | 15 | 44
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 Years) | 29 | 15 | 44
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 15 | 44
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Region was recorded for the total number of participants enrolled, not broken down into randomized groups.
  participants
    Turkey | 0 | 0 | 3
    United States | 0 | 0 | 10
    Italy | 0 | 0 | 2
    Mexico | 0 | 0 | 18
    Israel | 0 | 0 | 1
    Bulgaria | 0 | 0 | 2
    Serbia | 0 | 0 | 2
    Spain | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete 10 Meter Walk/Run[
Description: 10 Meter Walk/Run is a motor function test to measure the functional capability in patients with DMD.
Time Frame: Baseline, Week 24
Population: Summary aggregate results for all participants enrolled into Period 1 and with a score at Week 24
Measure: Median (Full Range); unit: seconds
Arm/Group | Period 1: MNK-1411 | Period 1: Placebo
Number analyzed (Participants) | 29 | 15
seconds
  at Baseline | 5.9 [4.7 to 22.3] | 7.8 [3.9 to 13.0]
  at Week 24: number analyzed (Participants) | 16 | 9
  at Week 24 | 5.4 [4.1 to 8.9] | 8.7 [3.3 to 18.3]

2. Secondary Outcome: North Star Ambulatory Assessment (NSAA) Score
Description: The NSAA is comprised of 17 items, each of which is graded using the standard scorecard. Each assessment is rated as 0 - unable to achieve independently, 1 - modified method but achieves goal independent of physical assistance from another, or 2 - normal with no obvious modification of activity. The subscale scores are summed for a total score ranging from 0 to 34. The higher the total score, the better the outcome.
Time Frame: Baseline, Week 24
Population: Summary aggregate results for all participants enrolled into Period 1 and with a score at Week 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Period 1: MNK-1411 | Period 1: Placebo
Number analyzed (Participants) | 29 | 15
score on a scale
  at Baseline | 17.9 (6.80) | 17.1 (6.40)
  at Week 24: number analyzed (Participants) | 17 | 9
  at Week 24 | 20.5 (7.94) | 16.6 (8.82)

3. Secondary Outcome: Time to Climb 4 Standardized Stairs
Description: Time to Climb 4 Standardized Stairs is a motor performance test
Time Frame: Baseline, Week 24
Population: Summary aggregate results for all participants enrolled into Period 1 and with a score at Week 24
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Period 1: MNK-1411 | Period 1: Placebo
Number analyzed (Participants) | 29 | 15
seconds
  at Baseline | 8.52 (8.88) | 8.47 (4.34)
  at Week 24: number analyzed (Participants) | 15 | 9
  at Week 24 | 4.71 (2.45) | 15.09 (13.84)

4. Secondary Outcome: Time to Stand From a Supine Position
Description: Time to stand from a supine position is a motor function test to measure the functional capability in subjects with DMD.
Time Frame: Baseline, Week 24
Population: Summary aggregate results for all participants who enrolled into Period 1 with a score for this measure at the given time point
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Period 1: MNK-1411 | Period 1: Placebo
Number analyzed (Participants) | 23 | 13
seconds
  at Baseline | 11.14 (9.08) | 15.03 (12.45)
  at Week 24: number analyzed (Participants) | 16 | 9
  at Week 24 | 7.65 (4.99) | 24.89 (26.48)

5. Secondary Outcome: Quantitative Muscle Testing Scores at Baseline
Description: Quantitative muscle testing measured strength-knee flexion and extension measured in Newtons, using a dynamometer
Time Frame: Baseline
Population: Summary aggregate results for all participants enrolled into Period 1 with a score at baseline.
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Period 1: MNK-1411 | Period 1: Placebo
Number analyzed (Participants) | 25 | 15
Newtons
  Knee flexion | 26.61 (14.17) | 29.87 (14.17)
  Knee extension | 28.99 (16.24) | 26.64 (15.27)

6. Secondary Outcome: Quantitative Muscle Testing Scores at Week 24
Description: Quantitative muscle testing measured strength-knee flexion and extension measured in Newtons, using a dynamometer
Time Frame: Week 24
Population: Summary aggregate results for all participants enrolled into Period 1 with a score at Week 24
Measure: Mean (Standard Deviation); unit: Newtons
Arm/Group | Period 1: MNK-1411 | Period 1: Placebo
Number analyzed (Participants) | 18 | 9
Newtons
  Knee flexion | 33.64 (1578) | 25.27 (13.35)
  Knee extension | 26.61 (14.17) | 29.87 (15.13)

7. Secondary Outcome: Summary of Adverse Events in the Blinded Treatment Period
Description: Clinically significant changes in vital signs, height, weight, immunogenicity and laboratory assessments were reported as adverse events (AEs)
Time Frame: within 28 weeks
Population: Summary aggregate results for all participants enrolled into Period 1
Measure: Count of Participants; unit: Participants
Arm/Group | Period 1: MNK-1411 | Period 1: Placebo
Number analyzed (Participants) | 29 | 15
Participants
  Exposed | 29 | 15
  Affected by serious adverse events | 0 | 1
  Affected by non-serious adverse events | 22 | 15
  Died from any cause | 0 | 0

8. Secondary Outcome: Summary of Adverse Events in the Open Label Period
Description: as for outcome 7
Time Frame: within 28 weeks
Population: Summary aggregate results for all participants enrolled into Period 2
Measure: Count of Participants; unit: Participants
Groups:
- Period 2: MNK-1411: All participants who received any dose of MNK-1411 in Period 2
Arm/Group | Period 2: MNK-1411
Number analyzed (Participants) | 24
Participants
  Exposed | 24
  Affected by serious adverse events | 2
  Affected by non-serious adverse events | 11
  Died from any cause | 0

ADVERSE EVENTS:
Time Frame: within 28 weeks
Description: Clinically significant changes in vital signs, height, weight, immunogenicity and laboratory assessment were reported as AEs
Groups:
- Period 2: MNK-1411: Participants receive MNK-1411 at a dosing volume appropriate to body weight during Period 2
Arm/Group | Period 1: MNK-1411 | Period 1: Placebo | Period 2: MNK-1411
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/15 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/15 | 2/24
Other Adverse Events (participants affected / at risk) | 22/29 | 15/15 | 11/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: MNK-1411 (N=29) | Period 1: Placebo (N=15) | Period 2: MNK-1411 (N=24)
Muscle disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
nary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: MNK-1411 (N=29) | Period 1: Placebo (N=15) | Period 2: MNK-1411 (N=24)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (2)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 1 (2) | 1 (2)
Face oedema (General disorders) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 4 (4) | 1 (1) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 4 (4) | 1 (1) | 2 (2)
Injection site irritation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site mass (General disorders) | 1 (1) | 3 (3) | 1 (1)
Injection site pain (General disorders) | 2 (2) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1)
Swelling face (General disorders) | 1 (1) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Separation anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 7 (9) | 0 (0) | 3 (3)
Nerve stimulation test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Congestive cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Cushingoid (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperphagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (4) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterobiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Scarlet fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT03400852/Prot_SAP_000.pdf